CLINICAL TRIAL: NCT04577833
Title: An Open-label, Randomized Study to Assess the Relative Bioavailability (BA) and Bioequivalence (BE) of Comparative Formulations of Niraparib and Abiraterone Acetate (AA) in Men With Prostate Cancer
Brief Title: A Study of Comparative Formulations of Niraparib and Abiraterone Acetate (AA) in Men With Prostate Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108783; 67652000PCR1001 (Other: Janssen Research & Development, LLC); 2019-000137-39 (EudraCT Number); 2023-508150-26-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2020-10-05; First posted 2020-10-08 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — niraparib; Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment Sequence ABD (Experimental): Participants will receive single doses of niraparib and abiraterone acetate (AA) using niraparib Formulation 1 as Treatment A in Treatment Period 1, followed by multiple doses of niraparib and AA using niraparib Formulation 2 as Treatment B in Treatment Period 2, followed by multiple doses of niraparib and AA using niraparib Formulation 4 as Treatment D in Treatment Period 3. From Period 2 onwards and during Extension and Long-term Extension Phases, all participants will continue to receive treatment with niraparib and AA-prednisone (AAP) or AAP alone.
  Interventions: Drug: Niraparib; Drug: Abiraterone Acetate (AA); Drug: Prednisone
- Treatment Sequence ADB (Experimental): Participants will receive Treatment A in Treatment Period 1 followed by Treatment D in Treatment Period 2, followed by Treatment B in Treatment Period 3. From Period 2 onwards and during Extension and Long-term Extension Phases, all participants will continue to receive treatment with niraparib and AAP or AAP alone.
  Interventions: Drug: Niraparib; Drug: Abiraterone Acetate (AA); Drug: Prednisone
- Treatment Sequence CBD (Experimental): Participants will receive single doses of niraparib and AA using niraparib Formulation 3 as Treatment C in Treatment Period 1, followed by Treatment B in Treatment Period 2, followed by Treatment D in Treatment Period 3. From Period 2 onwards and during Extension and Long-term Extension Phases, all participants will continue to receive treatment with niraparib and AAP or AAP alone.
  Interventions: Drug: Niraparib; Drug: Abiraterone Acetate (AA); Drug: Prednisone
- Treatment Sequence CDB (Experimental): Participants will receive Treatment C in Treatment Period 1, followed by Treatment D in Treatment Period 2, followed by Treatment B in Treatment Period 3. From Period 2 onwards and during Extension and Long-term Extension Phases, all participants will continue to receive treatment with niraparib and AAP or AAP alone.
  Interventions: Drug: Niraparib; Drug: Abiraterone Acetate (AA); Drug: Prednisone

INTERVENTIONS:
Drug: Niraparib — Niraparib will be administered orally.
Drug: Abiraterone Acetate (AA) — Abiraterone Acetate will be administered orally.
Drug: Prednisone — Prednisone will be administered orally.

SUMMARY:
The purpose of this study is to determine the relative bioavailability (rBA; Period 1) and bioequivalence (BE; Period 2 and 3) of various strengths and formulations of niraparib and abiraterone acetate (AA) at steady state under modified fasted conditions in participants with metastatic castration-resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
Niraparib is an orally available, highly selective poly (adenosine diphosphate [ADP]-ribose) polymerase (PARP) inhibitor, with potent activity against PARP-1 and PARP-2 deoxyribonucleic acid (DNA)-repair polymerases. AA is a pro-drug of abiraterone which selectively inhibits the enzyme 17 alpha-hydroxylase/C17,20-lyase (CYP17), that is found in the testes and adrenals (leading to systemic inhibition of testosterone production), as well as in prostate tissues and tumors. The rationale of the study is to investigate the various strengths and formulations of niraparib and AA plus prednisone or prednisolone (P) in metastatic castration resistant prostate cancer (mCRPC) participants with and without homologous recombination repair (HRR) gene alterations. In participants with metastatic prostate cancer, DNA-repair anomalies are found in approximately 15 percent (%) to 20% of tumors. This study consists 4 periods: screening phase (up to 21 days); treatment phase (up to 22 days); extension and long-term extension phases (from day 23 until discontinuation); and post-treatment follow up phase (end of treatment [EoT] visit within 30 days after the last dose of study treatment). Total duration of study is up to 1.4 years. Efficacy, safety, pharmacokinetics (PK), and biomarkers will be assessed at specified time points during this study. Participants safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Diagnosed with metastatic castration-resistant prostate cancer (mCRPC), who in the opinion of the investigator may benefit from treatment in this study
* Able to continue gonadotropin-releasing hormone analogues (GnRHa) therapy during the study if not surgically castrate (that is, participants who have not undergone bilateral orchiectomy)
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of less than or equal to (<=) 1
* Willing to provide a tumor sample (archival) for determination of homologous recombination repair (HRR) gene alteration status

Exclusion Criteria:

* Symptomatic brain metastases
* Prior disease progression during treatment with abiraterone acetate (AA) alone or when combined with a poly adenosine diphosphate (ADP)-ribose polymerase inhibitor (PARPi). Prior discontinuation of treatment with AA or PARPi due to AA- or PARPi related toxicity.
* History or current diagnosis of myelodysplastic syndrome (MDS)/ acute myeloid leukemia (AML)
* Known allergies, hypersensitivity, or intolerance to niraparib or AA or the corresponding excipients of niraparib/AA
* Any medical condition that would make prednisone/prednisolone use contraindicated

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Analyte Concentration at Steady State (Cmax,ss) of Niraparib and Abiraterone Acetate (AA) [Period 2 and Period 3] | Predose, up to 10 hour post dose
  Cmax,ss is defined as maximum observed analyte concentration at steady state.
Area Under the Plasma Concentration-time Curve from Time Zero to 24 Hours at Steady State (AUC [0-24h],ss) of Niraparib and AA (Period 2 and Period 3) | Predose, up to 24 hours post dose
  AUC (0-24h),ss is defined as area under the plasma concentration-time curve from time zero to 24 hours at steady state.
Ratio of Individual Cmax,ss Values Between Test and Reference Treatment (Period 2 and Period 3) | Predose, up to 10 hours post dose
  Ratio of individual Cmax,ss values between test and reference treatment will be assessed.
Ratio of individual AUC (0-24h),ss Values Between Test and Reference Treatment (Period 2 and Period 3) | Predose, up to 24 hours post dose
  Ratio of individual AUC (0-24h),ss values between test and reference treatment will be assessed.

SECONDARY OUTCOMES:
Maximum Observed Analyte Concentration at (Cmax) of Niraparib and AA (Period 1) | Predose, up to 72 hours post dose
  Cmax is defined as maximum observed analyte concentration.
Area Under the Plasma Concentration-time Curve from Time Zero to 72 Hours (AUC [0-72h]) of Niraparib and AA (Period 1) | Predose, up to 72 hours post dose
  AUC (0-72h) is defined as area under the plasma concentration-time curve from time zero to 72 hours post dosing.
Ratio of individual AUC (0-72h) Values Between Test and Reference Treatment (Period 1) | Predose, up to 72 hours post dose
  Ratio of individual AUC (0-72h) values between test and reference treatment will be assessed.
Serum Testosterone Level | Predose on Day -7, Day 11, Day 12 and Day 23
  Serum testosterone level will be assessed.
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | From study start until study completion (up to 3.1 years)
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with AEs by Severity | From study start until study completion (up to 3.1 years)
  Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death.
Number of Participants with Clinical Laboratory Abnormalities | From study start until study completion (up to 3.1 years)
  Number of participants with clinical laboratory abnormalities including hematology, serum chemistry and urinalysis will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (16):
- START Mountain Region, West Valley City, Utah, United States
- Belgium (2):
  - Universitair Ziekenhuis Gent, Ghent
  - GZA Ziekenhuizen- Campus St Augustinus, Wilrijk
- France (2):
  - Institut Bergonié, Centre de Lutte Contre le Cancer, Bordeaux
  - HIA Begin, Saint-Mandé
- Arensia Exploratory Medicine, Tbilisi, Georgia
- Arensia Exploratory Medicine, Chisinau, Moldova
- Erasmus MC, Rotterdam, Netherlands
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut Badawczy, Warsaw
- Spain (3):
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Hosp Univ Hm Sanchinarro, Madrid
  - Hosp Virgen de La Victoria, Málaga
- Karolinska Universitetssjukhuset Solna, Stockholm, Sweden
- ARENSIA Exploratory Medicine Unit, Kyiv, Ukraine
- Sir Bobby Robson Unit, Northern Centre for Cancer Care, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Yu A, Hazra A, Jiao JJ, Hellemans P, Mitselos A, Tian H, Ruixo JJP, Haddish-Berhane N, Ouellet D, Russu A. Demonstrating Bioequivalence for Two Dose Strengths of Niraparib and Abiraterone Acetate Dual-Action Tablets Versus Single Agents: Utility of Clinical Study Data Supplemented with Modeling and Simulation. Clin Pharmacokinet. 2024 Apr;63(4):511-527. doi: 10.1007/s40262-023-01340-5. Epub 2024 Mar 4. PMID 38436924